CLINICAL TRIAL: NCT04025775
Title: An Open-label, Two-centre, Randomised, 2-period Cross-over Study to Assess the Efficacy, Safety and Utility of Fully Closed-loop Insulin Delivery in Comparison With Standard Care, in Adults With Type 2 Diabetes Requiring Maintenance Dialysis
Brief Title: Closed-loop in Adults With T2D Requiring Dialysis
Acronym: AP-Renal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cambridge (Other)
Collaborators: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Principal Investigator, Dr Roman Hovorka, Professor of Metabolic Technology, University of Cambridge
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: AP-Renal
Record Dates: First submitted 2019-07-16; First posted 2019-07-19 (Actual); Last update posted 2022-05-17 (Actual); Status verified 2022-05

CONDITIONS: Type 2 Diabetes; End Stage Renal Disease
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Closed loop insulin delivery (Experimental): Unsupervised home use of day and night fully automated closed loop insulin delivery system (CamAPS HX) for 20 days
  The CamAPS HX closed-loop system comprises
  * Dana insulin pump (Diabecare, Sooil, Seoul, South Korea)
  * Dexcom G6 real-time CGM sensor (Dexcom, Northridge, CA, USA)
  * An Android smartphone hosting CamAPS HX Application with the Cambridge model predictive control algorithm and communicating wirelessly with the insulin pump
  * Glooko/Diasend cloud upload system to monitor CGM/insulin data.
  Interventions: Device: CamAPS HX Closed-loop
- Standard therapy (Active Comparator): Participants in the control arm will continue to follow their current diabetes management plan for the 20 day study period.Participants will be wear a masked continuous glucose monitoring (CGM) system during the 20 day study period.
  Interventions: Other: Multiple Daily Insulin Injections (Control)

INTERVENTIONS:
Device: CamAPS HX Closed-loop — The CamAPS HX closed-loop system comprises
  * Dana insulin pump (Diabecare, Sooil, Seoul, South Korea)
  * Dexcom G6 real-time CGM sensor (Dexcom, Northridge, CA, USA)
  * An Android smartphone hosting CamAPS HX Application with the Cambridge model predictive control algorithm and communicating wirelessly with the insulin pump
  * Glooko/Diasend cloud upload system to monitor CGM/insulin data.
  Arms: Closed loop insulin delivery
Other: Multiple Daily Insulin Injections (Control) — Multiple Daily Insulin Injections with masked Dexcom G6 CGM sensor (Dexcom, Northridge, CA, USA)
  Arms: Standard therapy

SUMMARY:
The main objective of this study is to determine the efficacy, safety and utility of fully automated closed-loop glucose control in the home setting over a 20 day period in adults with type 2 diabetes (T2D) requiring maintenance dialysis. This study builds on previous and on-going studies of closed-loop systems that have been performed in Cambridge in adults with type 1 diabetes in the home setting, and in adults with type 2 diabetes in the inpatient setting.

This is an open-label, two-centre, randomised, cross-over study, involving two home study periods during which glucose levels will be controlled either by a fully automated closed-loop system or by participants' usual insulin therapy in random order. Each treatment arm is 20 days long with a 2-4 week washout period between treatments. A total of up to 40 adults with T2D requiring maintenance dialysis will be recruited through outpatient clinics or the dialysis unit, to allow for 32 completed participants available for assessment.

Participants will receive appropriate training by the research team on the safe use of the study devices (insulin pump and continuous glucose monitoring (CGM) and closed-loop insulin delivery system). Participants in the control arm will continue with standard therapy and will wear a blinded CGM system.

The primary outcome is time spent with glucose levels in the target range between 5.6 and 10.0 mmol/L as recorded by CGM. Secondary outcomes are the time spent with glucose levels above and below target, as recorded by CGM, and other CGM-based metrics in addition to insulin requirements. Safety evaluation comprises the tabulation of severe hypoglycaemic episodes.

DETAILED DESCRIPTION:
Purpose of clinical trial To determine the efficacy, safety and utility of fully automated closed-loop insulin delivery in the home setting in adults with type 2 diabetes requiring maintenance dialysis.

Study objectives The study objective is to compare fully automated closed-loop insulin delivery with usual care in adults with type 2 diabetes requiring maintenance dialysis.

1. EFFICACY: The objective is to assess the ability of fully-automated closed-loop insulin delivery in maintaining CGM glucose levels within the target range from 5.6 to 10.0 mmol/l as compared to usual care in adults with type 2 diabetes requiring maintenance dialysis.
2. SAFETY: The objective is to evaluate the safety of fully automated closed-loop insulin delivery in terms of episodes and severity of hypoglycaemia, and nature and severity of other adverse events.
3. UTILITY: The objective is to determine the acceptability and duration of use of the closed-loop system.

Study design An open-label, two-centre, randomised, two-period crossover study comparing fully automated closed-loop insulin delivery with usual care in adults with type 2 diabetes requiring dialysis. Two intervention periods in the home setting will last 20 days each with a 2-4 week washout period. The order of the two interventions will be random.

Study endpoints The primary endpoint is the time spent in the target glucose range from 5.6 to 10.0 mmol/l based on CGM glucose levels during the 20 day home stay.

Other key endpoints:

* Time spent with sensor glucose above target (10.0 mmol/l)
* Time spent with sensor glucose <3.9 mmol/l
* Average of sensor glucose levels

Secondary endpoints include:

* Time spent with sensor glucose below target (5.6 mmol/l)
* Time spent with sensor glucose <3.0 mmol/l)
* Time spent with sensor glucose levels in significant hyperglycaemia (glucose levels > 20 mmol/l)
* Standard deviation and coefficient of variation of sensor glucose levels
* AUC of glucose below 3.5 mmol/l (63 mg/dl)
* Total daily insulin requirements
* Average inter-dialytic weight gain

Safety evaluation Assessment of frequency and severity of hypoglycaemic episodes and nature and severity of other adverse events.

Utility evaluation Assessment of the acceptability and duration of use of the closed-loop system.

Participating clinical centres

UK 1. Addenbrooke's Hospital, Cambridge University Hospitals NHS Foundation Trust, Cambridge,

Switzerland

1. Bern University Hospital, Bern

Sample size 32 adults completing the study. Recruitment will target up to 40 adults to allow for drop-outs.

Maximum duration of study for a participant 12 weeks

Recruitment Participants will be recruited through the adult diabetes outpatient clinics or dialysis units at participating centres.

Consent Written informed consent will be obtained from participants according to Research Ethics Committee (REC) requirements.

Screening and baseline assessment Eligible participants will undergo a baseline evaluation including medical (diabetes) history and current therapy.

Randomisation Eligible participants will be randomised in a 1:1 ratio using randomisation software to the use of fully automated closed-loop insulin delivery or to usual care for 20 days, with a 2-4 week washout period between the two interventions.

1. Closed loop arm Following randomisation, participants in the closed-loop group will receive training to cover key aspects of insulin pump use and CGM. Competency on the use of study devices will be evaluated Once competent in the use of the study pump and CGM, participants will receive training required for safe and effective use of the closed-loop system. During a 2-4 hour session participants will operate the system under the supervision of the clinical team. Competency on the use of closed-loop system will be evaluated. Thereafter, participants are expected to use closed-loop for 20 days without supervision or remote monitoring.

   All participants will be provided with 24 hour telephone helpline and will also be given written instructions about when to contact clinical team.
2. Standard therapy (control arm) Participants in the control group will continue with standard insulin therapy with blinded CGM for 20 days.

Study contacts Follow up contacts will be conducted within 24 hours of starting each treatment arm and then at weekly intervals thereafter.

End of study assessments Validated questionnaires evaluating the impact of the technology on diabetes management and quality of life will be completed. Participants will resume usual care.

Procedures for safety monitoring during trial Standard operating procedures for monitoring and reporting of all adverse events (AE) will be in place, including serious adverse events (SAE), serious adverse device effects (SADE).

A data safety and monitoring board (DSMB) will be informed of all serious adverse events and any unanticipated serious adverse device effects that occur during the study and will review compiled adverse event data at periodic intervals.

Criteria for withdrawal of patients on safety grounds

A participant may terminate participation in the study at any time without necessarily giving a reason and without any personal disadvantage. An investigator can stop the participation of a subject after consideration of the benefit/risk ratio. Possible reasons are:

1. Serious adverse events
2. Significant protocol violation or non-compliance
3. Failure to satisfy competency assessment
4. Decision by the investigator, or the Sponsor, that termination is in the participant's best medical interest
5. Pregnancy, planned pregnancy, or breast feeding
6. Allergic reaction to insulin

Efforts will be made to retain participants in follow up for the final primary outcome assessment even if the intervention is discontinued, unless the investigator believes that it will be harmful for the participant to continue in the trial.

ELIGIBILITY:
Inclusion Criteria:

* The subject is age 18 years or over
* Diagnosis of type 2 diabetes using standard diagnostic practice
* The subject requires maintenance dialysis
* The subject requires current treatment with subcutaneous insulin
* Screening HbA1c ≤ 11% (97mmol/mol) on analysis from local laboratory
* Subject is willing to perform regular finger-prick blood glucose monitoring
* The subject is literate in English (UK) or German (Switzerland)
* The subject is willing to wear study devices 24/7 during intervention arm and follow study specific instructions

Exclusion Criteria:

* Physical or psychological condition likely to interfere with the normal conduct of the study and interpretation of the study results as judged by the investigator
* Known or suspected allergy to insulin
* Lack of reliable telephone facility for contact
* Pregnancy, planned pregnancy, or breast feeding
* Severe visual impairment
* Severe hearing impairment
* Medically documented allergy towards the adhesive (glue) of plasters or unable to tolerate tape adhesive in the area of sensor placement
* Serious skin diseases located at places of the body, which potentially are possible to be used for localisation of the glucose sensor
* Illicit drugs abuse
* Prescription drugs abuse
* Alcohol abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Time in the target glucose range (5.6 to 10.0 mmol/l) | 20 day intervention period
  Percentage of time spent with sensor glucose readings in the target range from 5.6 to 10.0

SECONDARY OUTCOMES:
Time spent above target glucose (10.0 mmol/l) | 20 day intervention period
  Both armsPercentage of time spent with sensor glucose readings above target glucose (10.0 mmol/l)
Mean glucose | 20 day intervention period
  Mean sensor glucose level
Time spent in hypoglycaemia (<3.9 mmol/l) | 20 day intervention period
  Percentage of time spent with sensor glucose readings <3.9 mmol/l
Time spent below target glucose (5.6 mmol/l) | 20 day intervention period
  Percentage of time spent with sensor glucose readings below target glucose (5.6 mmol/l)
Standard deviation of glucose levels | 20 day intervention period
  Standard deviation of glucose levels
Coefficient of variation of glucose levels | 20 day intervention period
  Coefficient of variation of glucose levels
Time spent below <3.0 mmol/l | 20 day intervention period
  Percentage of time spent with sensor glucose readings <3.0 mmol/l
Time in significant hyperglycaemia (> 20 mmol/l) | 20 day intervention period
  Percentage of time with glucose levels in significant hyperglycaemia (> 20 mmol/l)
Total, basal and bolus insulin dose | 20 day intervention period
  Average daily total, basal and bolus insulin requirements
AUC of glucose below 3.5 mmol/l | 20 day intervention period
  Area under the curve of sensor glucose readings below 3.5mmol/l

OTHER OUTCOMES:
Number of episodes of severe hypoglycaemia | 20 day intervention period
  Safety evaluation
Number of subjects experiencing severe hypoglycaemia | 20 day intervention period
  Safety evaluation
Frequency and nature of other adverse events or serious adverse events | 20 day intervention period
  Safety evaluation
Percentage of time of closed-loop operation | 20 day intervention period
  Utility evaluation
Percentage of time of CGM availability | 20 day intervention period
  Utility evaluation
Average inter-dialytic weight gain | 20 day intervention period

CONTACTS AND LOCATIONS:
Overall Officials: Roman Hovorka, PhD, Study Director — University of Cambridge
Locations (2):
- Inselspital, Bern University Hospital, Bern, Switzerland
- Cambridge University Hospitals NHS Foundation Trust, Cambridge, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Fully anonymised data may be shared with third parties (EU or non-EU based) for the purposes of advancing management and treatment of diabetes.

REFERENCES:
- [Derived] Boughton CK, Tripyla A, Hartnell S, Daly A, Herzig D, Wilinska ME, Czerlau C, Fry A, Bally L, Hovorka R. Fully automated closed-loop glucose control compared with standard insulin therapy in adults with type 2 diabetes requiring dialysis: an open-label, randomized crossover trial. Nat Med. 2021 Aug;27(8):1471-1476. doi: 10.1038/s41591-021-01453-z. Epub 2021 Aug 4. PMID 34349267